CLINICAL TRIAL: NCT03900481
Title: Use of an Endoluminal-suturing Device for Endoscopic Gastric Reduction as an Aid for Class I Obesity, or Class II Obesity Without Comorbidity
Acronym: SLEEVE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Premature end of inclusion
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-18; 2019-A00261-56 (Other: ANSM)
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Bariatric Surgery; Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vertical gastric plication (Experimental): Vertical gastric plication ( without cutting gastric wall) is a novel surgical approach for reducing the stomach capacity. A transoral or endoluminal approach (i.e. a procedure that requires no incision, because access is granted through the mouth) offers some potential additional benefit to the patient, because the procedures continue to become more and more minimally invasive
  Interventions: Procedure: Vertical gastric plication

INTERVENTIONS:
Procedure: Vertical gastric plication — Vertical gastric plication ( without cutting gastric wall) is a novel surgical approach for reducing the stomach capacity. A transoral or endoluminal approach (i.e. a procedure that requires no incision, because access is granted through the mouth) offers some potential additional benefit to the patient, because the procedures continue to become more and more minimally invasive.

SUMMARY:
The primary objective is to measure the impact of this treatment for patients with obesity of class I, or class II without co-morbidity, assessed by excess weight loss (EWL)>25%. The secondary objectives are to measure total body weight loss >5%, BMI reduction, tolerance, complications related to this technique in this indication. This study is a prospective, pilot, bi-center safety and efficacy study. 30 patients will be enrolled between APHM, Marseille et CHU L'Archet Nice

DETAILED DESCRIPTION:
Surgery is currently the only effective treatment for morbid obesity and can be divided into restrictive surgeries (Sleeve gastrectomy), or malabsorptive surgery (Bypass surgery). The good medical practice guidelines recommend bariatric surgery for patients with body mass index (BMI) greater than 40 kg/m² without co-morbidities or between 35 and 40 kg/m² with co-morbidities (cardiovascular diseases, diabetes, sleep apnea, etc). Bariatric surgery is currently not an option for obese patients with a BMI between 30 and 35 kg/m² with or without comorbidities (Class I) or with a BMI between 35 and 40 kg/m² without comorbidity (Class II without comorbidity). Patients with obesity of class I, or class II without co-morbidity, currently have no possibility of interventional treatment other than nutritional therapy.

Vertical gastric plication ( without cutting gastric wall) is a novel surgical approach for reducing the stomach capacity. A transoral or endoluminal approach (i.e. a procedure that requires no incision, because access is granted through the mouth) offers some potential additional benefit to the patient, because the procedures continue to become more and more minimally invasive. Advances in endoluminal devices are now allowing clinicians the ability to begin exploring bariatric procedures performed via flexible endoscopy. Although these procedures may not be as effective as their surgical counterparts, these less-invasive options may relieve patients of the significant risks associated with surgery and might become part of the armamentarium of obesity management (5). Endomina (Endo Tools Therapeutics, Gosselies, Belgium) is a CE marked device that offers the possibilities of making transoral full thickness tissue apposition and may allow performing, via a transoral route, large plications with tight serosa to serosa apposition.

The investigators wish to carry out a bi-centric pilot study (Marseille, Nice) which will validate the effectiveness (in terms of excess weight loss and total body weight loss) of this new endoscopic technique for patients previously excluded from any surgical management of their obesity (class I, or class II without comorbidity). The primary objective is to measure the impact of this treatment for patients with obesity of class I, or class II without co-morbidity, assessed by excess weight loss (EWL)>25%. The secondary objectives are to measure total body weight loss >5%, BMI reduction, tolerance, complications related to this technique in this indication. This study is a prospective, pilot, bi-center safety and efficacy study. 30 patients will be enrolled between APHM, Marseille et CHU L'Archet Nice

ELIGIBILITY:
Inclusion Criteria:

* 18 years ≤ age ≤ 65 years
* Class I obesity (30 <BMI <35 kg / m²) or Class II without comorbidity (35 <BMI <40 kg / m²)

Exclusion Criteria:

* Achalasia or other disturbance of motility of the esophagus;
* severe esophagitis;
* Peptic ulcer disease;* uncontrolled diabetes
* Weight loss> 5% of the total weight over the last 6 months;
* Gastrointestinal stenosis or obstruction;
* Pregnancy, breastfeeding, or desire for pregnancy in the next 18 months;
* Previous bariatric surgery, balloon or other endoscopic therapy of obesity;
* Gastric surgery scheduled within 60 days of surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
Assessment of the excess weight loss | 12 months
  Measure the impact of this treatment for patients with obesity of class I, or class II without co-morbidity, assessed by excess weight loss (EWL)>25%

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Garrido-Pradalie, Study Director — Assistance Publique- Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France